CLINICAL TRIAL: NCT04291001
Title: A Pilot Prospective, Randomized Pharmacodynamic Study With Assessment of Ulipristal Acetate on Ovarian Activity Following Quickstart of the Etonogestrel Contraceptive Implant
Brief Title: Ovarian Function With ENG Implant and UPA Use
Status: Completed | Phase: Early Phase 1 | Type: Interventional
Sponsor: University of Utah (Other)
Collaborators: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Other
Other Study IDs: 129999
Record Dates: First submitted 2020-02-27; First posted 2020-03-02 (Actual); Results first posted 2024-07-12 (Actual); Last update posted 2024-07-12 (Actual); Status verified 2024-07

CONDITIONS: Contraception
Keywords: emergency contraception; contraceptive implant; ovulation
MeSH Terms: interventions — Electronystagmography; ulipristal acetate

STUDY DESIGN:
Intervention Model Description: Randomization scheme: block randomization with block size of 4
  Blinding protocol: This study will not be blinded as a pilot. The feasibility of the study, including clinic space limitations and provider time, relies on the same healthcare provider for implant insertion and ultrasound in many patients. All statistical analyses will be blinded to the statistician.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: Yes

ARMS (2):
- ENG Implant alone (Active Comparator): Participants will receive a contraceptive implant in the setting of a dominant follicle to assess ovulation incidence and timing following insertion.
  Interventions: Device: ENG implant
- ENG Implant plus oral UPA (Active Comparator): Participants will receive a contraceptive implant and oral UPA the same day in the setting of a dominant follicle to assess ovulation incidence and timing following insertion.
  Interventions: Device: ENG implant; Drug: oral ulipristal acetate

INTERVENTIONS:
Device: ENG implant — This is an FDA-approved contraceptive device
  Other Names: Nexplanon
Drug: oral ulipristal acetate — This is an FDA-approved oral emergency contraceptive
  Other Names: Ella
  Arms: ENG Implant plus oral UPA

SUMMARY:
Same day initiation of the etonogestrel (ENG) implant and oral ulipristal acetate (UPA) would overcome contraceptive access barriers to people capable of pregnancy with recent unprotected intercourse to ongoing contraception. Current clinical guidelines recommend delaying implant initiation for at least 1 week following UPA, as well as waiting 7 days before relying on the implant for contraception after initiation alone. This pilot will assess the effects of the implant alone and the implant inserted with same-day as UPA usage on ovarian activity. A total of 40 people capable of pregnancy desiring the implant, who are not at risk for pregnancy during the study timeline, will be recruited. Participants will be randomized to implant alone or same-day implant + oral UPA. Participants will have daily ultrasounds and blood draws to assess timing of ovulation for 1 week and then an exit visit at 14 days after randomization. The primary outcome is the incidence of ovulation in the 2 randomized treatment groups. Participants may continue the implant after the study per FDA guidelines and rely on it for contraception after the study is completed.

DETAILED DESCRIPTION:
Primary Objectives:

1. To determine point estimates for the incidence of ovulation within five days of oral ulipristal acetate (UPA) administration with same day etonogestrel (ENG) implant insertion in the presence of a dominant follicle.
2. To determine point estimates for the incidence of ovulation within five days of etonogestrel (ENG) implant insertion alone in the presence of a dominant follicle.

   .

Clinical hypotheses:

• Combined oral UPA administration with same day ENG implant insertion will interfere with UPA's effect in delaying ovulation as occurs with oral progestogens given within 1-2 days of UPA.

Study Design: Pilot randomized, single site clinical trial with blinded analysis

Participant recruitment and study site: The investigators will recruit participants interested in using the ENG contraceptive implant but not currently at risk for pregnancy from Planned Parenthood Association of Utah clinics, University of Utah Hospital and Community clinics, and through targeted social media ads. All study procedures will occur at the University of Utah Hospital Outpatient OBGYN Clinic or at the University Center for Reproductive Medicine clinic.

Sample size: This is a pilot proposal to recruit a total of 40 participants across 2 study arms: (1) ENG implant only (n=20) and (2) UPA + same day ENG implant insertion (n=20). The investigators null hypotheses are:

1. ENG implant along with UPA administration in the presence of a dominant ovarian follicle will not change the expected 97% ovulation suppression within 5 days of UPA use.
2. ENG implant insertion alone in the presence of a dominant ovarian follicle will not sufficiently interrupt ovulation.

Randomization scheme: block randomization with block size of 4

Blinding protocol: This study will not be blinded as a pilot. The feasibility of the study, including clinic space limitations and provider time, relies on the same healthcare provider for implant insertion and ultrasound in many patients. All statistical analyses will be blinded to the statistician.

Participant procedures:

Screening Visit (Screening Visit 1): Subjects will be screened for eligibility and interest in the study. Each subject will have the study explained and, if participation is desired, informed consent documents will be signed prior to any study procedures. The screening visit will include: review of medical, surgical and social history, medications, menstrual dating, sexual history and contraceptive use, physical exam, including breast and pelvic, pregnancy test and a transvaginal ultrasound to ensure ability to document ovarian follicular activity in the treatment cycle.

Progesterone Visit (Screening Visit 2): This brief visit will occur on days 20-24 of the menstrual cycle and may be combined with the screening visit (Visit 1) if the time-frame is met. This visit will include a review of any interim changes (if completed separate from the screening visit) in history, medications, pregnancy risk/contraception, and a serum progesterone level will be drawn. The participants will notify the study coordinator of the 1st day of their next menses.

Ovarian monitoring (Screening Visits 3-7 +/- 2 visits): Participants will undergo transvaginal ultrasound evaluation of their ovaries three times a week starting on cycle day #7 (+/- 2 days). If/ When investigators identify a lead follicle with a mean diameter of >13mm in at least 2 dimensions, study follow-up will switch to daily monitoring.

Treatment Day #1 (Treatment Visit #1): Once a lead follicle (>14mm) is identified then participants will be randomized to one of two treatment groups:

1. ENG implant insertion
2. UPA 30mg PO tablet and same-day ENG implant insertion Assigned treatment will be administered (UPA and/or ENG implant insertion). Study team will obtain serum progesterone, LH levels, and estradiol levels.

Treatment Days #2-8 (Treatment Visits #2-8): Participants will follow up daily for Days 2-8. Each day investigators will obtain transvaginal ultrasound measurement of ovarian follicle size, serum progesterone, LH levels, and estradiol levels. Daily transvaginal ultrasounds will continue until either follicle rupture is documented, the follicle is <12 mm on two consecutive visits, or Day 8 ultrasound occurs (7 days after implant insertion), whichever occurs first.

Treatment Day #14 (Exit Visit): Repeat ultrasound will occur on Day 14 following ENG implant insertion, and this will be the exit visit.

Data collection: Source documents for each participant and visit number will be completed by the study personnel at the time of the visit. Form development, data collection, and data management will occur in RedCAP, secure web platform for building and managing online databases and surveys. Source documents maintained in individual participant binders.

Assessing and reporting adverse events: The reporting period for AEs is the period immediately following the subject signing the informed consent through the 30 days following the final study visit. Each visit will include assessment of how the participant felt since the last visit, review of adverse event reports, implant insertion site reactions, lab results, and vital signs and physical exam findings. AEs will not be reported for screen failures unless a SAE is experienced during screening. For all AEs, the investigator will pursue and obtain information adequate to determine the outcome of the AE and to assess whether it met criteria for a SAE. Participants who have ongoing AEs or SAEs will be followed until resolution or stabilization or referred for additional care. AEs will be documented both on source documents and in the clinical database with SAEs reported per IRB guidelines. Participants will be provided instructions for contacting the study site to report any untoward medical occurrences. With permission from the participant, whenever possible records from all non-study medical providers related to medical occurrences will be obtained for review. AEs and SAEs will be reviewed by the Data Safety Monitoring Board.

Statistical Analyses:

The investigator and study team will be responsible for analyzing the study data. The official clinical database in RedCAP will not be analyzed until medical/scientific review has been completed, protocol violators have been identified (if appropriate), and data has been declared complete.

Variables/Time Points of Interest The primary outcome is delay in rupture of the dominant follicle by 5 days (yes/no) between group 1 (ENG implant alone) and group 2 (UPA with same day ENG implant). If the date of follicle rupture was unclear by ultrasound alone, investigators will utilize serum hormone levels to adjudicate day of rupture. These measures include day of follicle collapse, day and value of highest LH, day and value of highest progesterone level. Investigators will use an estradiol level of >100pg/ml to confirm the enlarged follicle is the dominant follicle on the treatment day.

Statistical Methods The primary and secondary dichotomous outcome measures of ovulation by 5 days will be assessed by Wilcoxon sign rank test and demographic will be analyzed using descriptive statistics.

Power/Sample Size:

The investigator and study team will be responsible for analyzing the study data. The official clinical database in RedCAP will not be analyzed until medical/scientific review has been completed, protocol violators have been identified (if appropriate), and data has been declared complete.

Variables/Time Points of Interest The primary outcome is delay in rupture of the dominant follicle by 5 days (yes/no) between group 1 (ENG implant alone) and group 2 (UPA with same day ENG implant). If the date of follicle rupture was unclear by ultrasound alone, investigators will utilize serum hormone levels to adjudicate day of rupture. These measures include day of follicle collapse, day and value of highest LH, day and value of highest progesterone level. Investigators will use an estradiol level of >100pg/ml to confirm the enlarged follicle is the dominant follicle on the treatment day.

This is a pilot study to obtain point estimates for future study proposals. Current data on ovulatory function with mid-cycle implant insertion or the pharmacodynamics interactions between same day UPA and ENG are lacking.

Should data show that ovulation occurs <15% within 5 days of combined UPA use and ENG implant initiation, investigators will pursue an adequately powered study assessing ovulation delay with UPA only vs. UPA with ENG implant initiation. This finding would show that UPA's relationship with the ENG implant may be different than what has been found with oral progestogens. If ovulation occurs 15% in the first 5 days with combined use of these medications, this would support the current practice of delaying implant insertion after UPA administration.

Should data show that the ENG implant insertion alone in the presence of a dominant follicle delays or stops ovulation >44% (the ovulation suppression of oral LNG EC), investigators will pursue an adequately powered study assessing the ENG implant alone for EC. If ovulation occurs >15%, this would support continuation of the practice of using a backup method when an implant is inserted after the first 7 days of the menstrual cycle.

These pre-specified criteria to judge if and how to proceed are consistent with CONSORT guidelines for randomized pilot and feasibility trials.[11]

ELIGIBILITY:
Inclusion Criteria:

* Healthy females, age 18-35
* Fluent in English
* BMI < 30 kg/m2
* No known contraindication to either the ENG contraceptive implant or Ulipristal Acetate (UPA) using the CDC Medical Eligibility Criteria for Contraceptive Use 2016
* Not current pregnant and not at risk of pregnancy (defined as not having penile-vaginal intercourse or using a non-hormonal method of contraception such as a barrier method, condoms, diaphragm, or cervical cap, a copper IUD, or permanent contraception)
* Know the date of last menstrual period
* Have a regular menstrual cycle (24-35 days)
* Be willing to comply with all study requirements
* Be willing to avoid pregnancy for the duration of the study

Exclusion Criteria:

* Currently pregnancy or breastfeeding
* Use of hormonal contraception or exogenous hormones (estrogen, progestogen, or HCG) in the last month (or past 6 months for depo medroxyprogesterone acetate) or planned use of such during the study
* Vaginal bleeding of unknown etiology
* Allergy to UPA or ENG
* Regular or planned use of glucocorticoids during the study
* Current or planned use of any medication that potentially interacts with UPA or ENG

Ages: 18 Years to 35 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 40 (Actual)
Dates: Start 2020-09-04 (Actual); Primary Completion 2022-10-10 (Actual); Study Completion 2024-01-12 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Lori Gawron, MD, Principal Investigator — University of Utah
Locations (1):
- University of Utah, Salt Lake City, Utah, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- ENG Implant Alone: Women will receive a contraceptive implant in the setting of a dominant follicle to assess ovulation incidence and timing following insertion.
  ENG implant: This is an FDA-approved contraceptive device
- ENG Implant Plus Oral UPA: Women will receive a contraceptive implant and oral UPA the same day in the setting of a dominant follicle to assess ovulation incidence and timing following insertion.
  ENG implant: This is an FDA-approved contraceptive device
  oral ulipristal acetate: This is an FDA-approved oral emergency contraceptive
Period: Overall Study
Arm/Group | ENG Implant Alone | ENG Implant Plus Oral UPA
Started | 20 | 20
Completed | 20 | 19
Not Completed | 0 | 1

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | ENG Implant Alone | ENG Implant Plus Oral UPA | Total
Number analyzed (Participants) | 20 | 20 | 40
Age, Continuous [Mean (Standard Deviation); unit: years] | 23.2 (3.9) | 24.3 (3.5) | 23.7 (3.7)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 20 | 20 | 40
  Male | 0 | 0 | 0
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 4
  Not Hispanic or Latino | 18 | 18 | 36
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 1 | 0 | 1
  Asian | 0 | 1 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 18 | 19 | 37
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 1 | 0 | 1
Region of Enrollment [Number; unit: participants]
  United States | 20 | 20 | 40
BMI [Mean (Standard Deviation); unit: kg/m^2] | 24.2 (2.7) | 23.7 (3.1) | 24.0 (2.9)

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants With Ovulation With Implant-alone
Description: Ovulation will be monitored by ultrasound and serum LH and progesterone levels
Time Frame: 5 days
Population: Outcome Measure was pre-specified to assess "ENG Implant Alone"
Measure: Count of Participants; unit: Participants
Groups:
- ENG Implant Plus Oral UPA: ParticipantsUPA the same day in the setting of a dominant follicle to assess ovulation incidence and timing following insertion.
  ENG implant: This is an FDA-approved contraceptive device
  oral ulipristal acetate: This is an FDA-approved oral emergency contraceptive
Arm/Group | ENG Implant Alone | ENG Implant Plus Oral UPA
Number analyzed (Participants) | 20 | 0
Participants | 7 | 0

2. Primary Outcome: Number of Participants With Ovulation With Implant and Same Day UPA
Description: Ovulation will be monitored by ultrasound and serum LH and progesterone levels
Time Frame: 5 days
Population: Outcome Measure was pre-specified to assess "ENG Implant plus oral UPA"
Measure: Count of Participants; unit: Participants
Arm/Group | ENG Implant Alone | ENG Implant Plus Oral UPA
Number analyzed (Participants) | 0 | 19
Participants | 0 | 13

ADVERSE EVENTS:
Time Frame: 30 days after final study visit, up to 44 days
Arm/Group | ENG Implant Alone | ENG Implant Plus Oral UPA
All-Cause Mortality (participants affected / at risk) | 0/20 | 0/20
Serious Adverse Events (participants affected / at risk) | 0/20 | 0/20
Other Adverse Events (participants affected / at risk) | 0/20 | 1/20
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | ENG Implant Alone (N=20) | ENG Implant Plus Oral UPA (N=20)
Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) — Participant requested removal of ENG implant on day 2 due to pain in left arm insertion site. Pain resolved after removal.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2024-01-12): https://cdn.clinicaltrials.gov/large-docs/01/NCT04291001/Prot_SAP_000.pdf